CLINICAL TRIAL: NCT01336075
Title: Atrial Fibrillation: Ablation or Surgical Treatment II: FAST II A Randomized Study Comparing Non-pharmacologic Therapy in Patients With Drug-refractory Atrial Fibrillation Referred for a First Time Invasive Treatment.
Brief Title: Atrial Fibrillation: Ablation or Surgical Treatment II: FAST II
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Too few participants
Sponsor: Aalborg University Hospital (Other)
Collaborators: St. Antonius Hospital (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Henrik Vadmann, MD, Ph.d student., MD, Ph.D. student, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FAST II
Record Dates: First submitted 2011-04-13; First posted 2011-04-15 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: Paroxysmal Atrial Fibrillation.
Keywords: Percutaneous radiofrequency catheter ablation; Mini invasive thoracoscopic radiofrequency ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation; Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mini invasive thoracoscopic radiofrequency ablation (Active Comparator): Video-assisted thoracoscopic radiofrequency ablation
  Interventions: Procedure: Mini invasive thoracoscopic radiofrequency ablation
- Percutaneous ablation (Active Comparator): Percutaneous radiofrequency catheter ablation
  Interventions: Procedure: Percutaneous radiofrequency catheter ablation

INTERVENTIONS:
Procedure: Percutaneous radiofrequency catheter ablation — Percutaneous radiofrequency catheter ablation around the rights and lefts pulmonary veins, with complete circumferential ablation.
  Other Names: Radiofrequency ablation; Catheter ablation; Atrial fibrillation ablation
  Arms: Percutaneous ablation
Procedure: Mini invasive thoracoscopic radiofrequency ablation — Video-assisted thoracoscopic approach for electrical isolation of the pulmonary veins bilaterally and left atrial appendage excision or exclusion.
  Other Names: Mini invasive mini maze
  Arms: Mini invasive thoracoscopic radiofrequency ablation

SUMMARY:
The purpose of this study is to compare two invasive treatments of symptomatic paroxysmal atrial fibrillation: Percutaneous radiofrequency catheter ablation and mini invasive thoracoscopic radiofrequency ablation in patients referred for a first time invasive treatment for atrial fibrillation.

The hypothesis is, that mini invasive thoracoscopic radiofrequency ablation as a first time invasive treatment is more effective compared to a percutaneous catheter based technique in patients with symptomatic paroxysmal atrial fibrillation refractory or intolerant to at least one antiarrhythmic drug.

DETAILED DESCRIPTION:
Atrial fibrillation is characterized by disorganized, rapid, and irregular contraction of the atria. Its effects on hemodynamic and thromboembolic events result in significant morbidity, mortality, impaired quality of life, hospitalizations, and health-cost.

It is the most common sustained cardiac arrhythmia. Over six million Europeans suffer from this arrhythmia. The prevalence is estimated to at least double in the next 50 years and is probably underestimated due to asymptomatic atrial fibrillation. The prevalence increases with age and affects men more often.

Atrial fibrillation is treated medically with varying results and there are no definitive long term curative treatments. The main goal aims at reducing symptoms and preventing disabling complications. Treatment normally includes antithrombotic, rhythm, and/or rate management, New non-pharmacological interventions have evolved over the last decades in order to prevent paroxysmal atrial fibrillation and/or reduce symptoms. The main focus of non-pharmacological intervention has been on percutaneous radiofrequency catheter ablation and surgical maze ablation. Both approaches aim at minimizing the impact of "triggers" from the pulmonary veins by electrical isolation of the veins.

Studies comparing antiarrhythmic drug and radiofrequency ablation indicate that radiofrequency ablation has a higher efficacy rate, a lower rate of complications, and in selected patients radiofrequency ablation reduced the risk of atrial fibrillation recurrence after one year by 65 % compared with antiarrhythmic drug. In a recently published paper the success rate after a mean of 1.3 radiofrequency ablation procedures per patient varied from 57.7% to 75.4% with higher success rates in patients with paroxysmal atrial fibrillation as compared to persistent/permanent atrial fibrillation.

European Society of Cardiology recommends that radiofrequency ablation is reserved for patients who remain symptomatic despite optimal therapy and failed at least one antiarrhythmic drug.

Dr. James Cox introduced the Cox-maze surgical operation for atrial fibrillation in 1987, later modified to Cox-maze III also known as the "cut and sew" maze. It is highly successful in restoring sinus rhythm, with 90-96 % being free from atrial fibrillation at a mean follow-up of 5.4 years. Due to its complexity and technical difficulty the procedure has not been widely adopted. Mini invasive procedures for pulmonary vein isolation have been developed and can now be performed either through mini thoracotomies or using totally thoracoscopic approach. These procedures also hold the advantage of left atrial appendage excision or exclusion. The thoracoscopic maze ablation has shown promising results in small studies in patients with recurrence of atrial fibrillation after earlier catheter based radiofrequency ablation, after a mean follow-up of 11 months 84 % of the patients remain in sinus rhythm. However long-term results are still unknown. The procedure still needs to be compared head to head with catheter based radiofrequency ablation before it should be offered as a standard treatment of atrial fibrillation.

The rationale for eliminating atrial fibrillation with radiofrequency ablation include a potential improvement in quality of life, decreased stroke risk, decreased heart failure risk and improved survival.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent symptomatic paroxysmal atrial fibrillation
* Previously failed one or more antiarrhythmic or beta-blocker medication (treatment > 30 days) or if any contraindications against treatment with these drug.
* Patient is willing and able to attend the scheduled follow-up visits
* Signed informed consent

Exclusion Criteria:

* Persistent or permanent atrial fibrillation
* Previously atrial fibrillation ablation procedure
* Atrial fibrillation secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause
* Severe underlying heart disease (congenital heart disease, significant valvular disease, cardiomyopathy with LVEF < 35 %, angina pectoris/ ischemic heart disease).
* Severe enlargement of left atrium (> 45mm)
* Patient with pacemaker
* Failure to obtain informed consent
* Pregnant or breastfeeding women.
* Patient unable to undergo TEE or with documented left atrial thrombus
* Patients with co-morbid conditions who, in the opinion of the investigator, constitute increased risk of general anesthesia or port access, e.g. pleural fibrosis, chronic obstructive pulmonary disease (FEV1 < 1.5 L/s).
* Known internal carotid artery stenosis (> 80 %).
* Patients, who are enrolled in another clinical trial
* Life expectancy less than one year
* Previously TIA/stroke

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Freedom from atrial fibrillation with or without antiarrhythmic drug. | 12 month follow-up
  Determined by seven days Holter monitoring, ECG, and patient interviews. An episode of atrial fibrillation/flutter/tachycardia is defined as more than 30 seconds of atrial fibrillation observed on Holter monitoring/telemetry or ECG

SECONDARY OUTCOMES:
Quality of life | 12 month follow-up
  Comparison of quality of life before ablation and at follow-up, by 4 different quality of life questionnaires AFEQT, AF-QoL-18, GAD-7 and PHQ-9.
Procedural complications | 12 month follow-up
  Thromboembolic events (TIA,Stroke), Mortality, Tamponade, need for thoracotomy, bleeding, infection, esophageal fistula, embolic events, death , pneumothorax and hemothorax.
Health economics (cost-effectiveness analysis) | 12 month follow-up
Reduction in atrial fibrillation burden | 12 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Vadmann, MD, Principal Investigator — Aalborg University Hospital; Sam Riahi, MD, PhD, Principal Investigator — Aalborg University Hospital; Jan Jesper Andreasen, MD, PhD, Principal Investigator — Aalborg University Hospital; Søren Hjortshøj, MD, PhD, Principal Investigator — Aalborg University Hospital; Alaaddin Yilmaz, MD, Principal Investigator — St. Antonius Hospital; Lucas Boersma, MD, PhD, Principal Investigator — St. Antonius Hospital; Axel Brandes, MD, FESC, Principal Investigator — Odense Universityhospital; Peter Pallesen, MD, Principal Investigator — Odense Universityhospital
Locations (3):
- Denmark (2):
  - Dept of Cardiothoracic surgery and Dept of Cardiology, Aalborg Hospital, Aalborg
  - Odense Universityhospital, Odense
- St. Antonius Hospital, Nieuwegein, Netherlands

REFERENCES:
- [Background] Camm AJ, Kirchhof P, Lip GY, Schotten U, Savelieva I, Ernst S, Van Gelder IC, Al-Attar N, Hindricks G, Prendergast B, Heidbuchel H, Alfieri O, Angelini A, Atar D, Colonna P, De Caterina R, De Sutter J, Goette A, Gorenek B, Heldal M, Hohloser SH, Kolh P, Le Heuzey JY, Ponikowski P, Rutten FH; ESC Committee for Practice Guidelines. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). Europace. 2010 Oct;12(10):1360-420. doi: 10.1093/europace/euq350. No abstract available. PMID 20876603
- [Background] Yilmaz A, Geuzebroek GS, Van Putte BP, Boersma LV, Sonker U, De Bakker JM, Van Boven WJ. Completely thoracoscopic pulmonary vein isolation with ganglionic plexus ablation and left atrial appendage amputation for treatment of atrial fibrillation. Eur J Cardiothorac Surg. 2010 Sep;38(3):356-60. doi: 10.1016/j.ejcts.2010.01.058. Epub 2010 Mar 12. PMID 20227287
- [Background] Nair GM, Nery PB, Diwakaramenon S, Healey JS, Connolly SJ, Morillo CA. A systematic review of randomized trials comparing radiofrequency ablation with antiarrhythmic medications in patients with atrial fibrillation. J Cardiovasc Electrophysiol. 2009 Feb;20(2):138-44. doi: 10.1111/j.1540-8167.2008.01285.x. Epub 2008 Sep 3. PMID 18775040
- [Background] Lafuente-Lafuente C, Mouly S, Longas-Tejero MA, Bergmann JF. Antiarrhythmics for maintaining sinus rhythm after cardioversion of atrial fibrillation. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD005049. doi: 10.1002/14651858.CD005049.pub2. PMID 17943835
- [Background] Schilling RJ. Cardioversion of atrial fibrillation: the use of antiarrhythmic drugs. Heart. 2010 Mar;96(5):333-8. doi: 10.1136/hrt.2008.155812. Epub 2009 Nov 11. PMID 19910286
- [Background] Calkins H, Reynolds MR, Spector P, Sondhi M, Xu Y, Martin A, Williams CJ, Sledge I. Treatment of atrial fibrillation with antiarrhythmic drugs or radiofrequency ablation: two systematic literature reviews and meta-analyses. Circ Arrhythm Electrophysiol. 2009 Aug;2(4):349-61. doi: 10.1161/CIRCEP.108.824789. Epub 2009 Jun 2. PMID 19808490
- [Background] Cappato R, Calkins H, Chen SA, Davies W, Iesaka Y, Kalman J, Kim YH, Klein G, Natale A, Packer D, Skanes A, Ambrogi F, Biganzoli E. Updated worldwide survey on the methods, efficacy, and safety of catheter ablation for human atrial fibrillation. Circ Arrhythm Electrophysiol. 2010 Feb;3(1):32-8. doi: 10.1161/CIRCEP.109.859116. Epub 2009 Dec 7. PMID 19995881
- [Background] Cox JL. Cardiac surgery for arrhythmias. J Cardiovasc Electrophysiol. 2004 Feb;15(2):250-62. doi: 10.1046/j.1540-8167.2004.03656.x. PMID 15028063
- [Background] Gaynor SL, Diodato MD, Prasad SM, Ishii Y, Schuessler RB, Bailey MS, Damiano NR, Bloch JB, Moon MR, Damiano RJ Jr. A prospective, single-center clinical trial of a modified Cox maze procedure with bipolar radiofrequency ablation. J Thorac Cardiovasc Surg. 2004 Oct;128(4):535-42. doi: 10.1016/j.jtcvs.2004.02.044. PMID 15457154
- [Background] Shen J, Bailey M, Damiano RJ Jr. Surgery for Lone Atrial Fibrillation: Present State-of-the-Art. Innovations (Phila). 2009 Oct;4(5):248-255. doi: 10.1097/IMI.0b013e3181bb370f. PMID 20473355
- [Derived] Sindby JE, Vadmann H, Lundbye-Christensen S, Riahi S, Hjortshoj S, Boersma LVA, Andreasen JJ. Percutaneous versus thoracoscopic ablation of symptomatic paroxysmal atrial fibrillation: a randomised controlled trial - the FAST II study. J Cardiothorac Surg. 2018 Oct 3;13(1):101. doi: 10.1186/s13019-018-0792-8. PMID 30285795